CLINICAL TRIAL: NCT01263210
Title: Conjugate Pneumococcal Vaccination - a Randomized Study in Young Otitis-prone Children
Brief Title: Pneumococcal Vaccination of Otitis-prone Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Financial support was provided by the Swedish Association of Local Authorities and Regions. The vaccine was kindly supplied by Wyeth Lederle. (Unknown)
Responsible Party: Marie Gisselsson Solén, ENT Department, Lund University Hospital, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LU62601
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-12

CONDITIONS: Recurrent Acute Otitis Media
Keywords: Recurrent acute otitis media; Conjugate pneumococcal vaccine; Ventilation tube treatment; Nasopharyngeal flora
MeSH Terms: conditions — Otitis Media | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pneumococcal vaccine (Active Comparator): Half of the children were randomized to receive heptavalent pneumococcal conjugate vaccine (before this vaccine was included in the national immunization programme).
  Interventions: Biological: Prevenar
- Control (No Intervention): Half of the children were randomized to no vaccination and functioned as controls.

INTERVENTIONS:
Biological: Prevenar
  Arms: Pneumococcal vaccine

SUMMARY:
Acute otitis media (AOM) is a common childhood disease, which becomes recurrent in 15-20% of the cases. Streptococcus pneumoniae is one of the leading causative agents, and a small reduction in the number of AOM episodes has been noted in unselected child cohorts after vaccination with conjugate heptavalent pneumococcal vaccine. This study was performed in order to investigate whether vaccination could reduce the number of AOM episodes in very young, otitis-prone children.

DETAILED DESCRIPTION:
Ninetysix children (46 vaccinated, 50 not) with an onset of AOM before six months of age, implying a high risk for developing rAOM, were recruited between 2003 and 2007. They were closely followed with clinical visits and nasopharyngeal cultures until the age of two years.

ELIGIBILITY:
Inclusion Criteria: First episode of acute otitis media before 6 months of age and verified by an otorhinolaryngologist.

-

Exclusion Criteria: Allergy to the vaccine, anatomical abnormality (eg cleft palate), chromosomal abnormality, immune deficiency, prematurity, prior administration of gammaglobulin or pneumococcal vaccine and a history of idiopathic thrombocytopenic purpura.

-

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2003-03; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Possible reduction of the number of acute otitis media episodes after conjugate pneumococcal vaccination in young otitis-prone children | 2 years
  Children with an acute otitis media onset before 6 months of age, implying an 80% risk for developing recurrent acute otitis media, were allocated to vaccination with heptavalent conjugate pneumococcal vaccine or to no vaccination. The number of acute otitis media episodes before two years of age in each group were recorded.

SECONDARY OUTCOMES:
Nasopharyngeal carriage in young otitis-prone children | 3 years
  The children in the vaccination study described above, had nasopharyngeal samples taken very frequently (every other month during the first year in the study, and at every suspected new episode of acute otitis media). The cultures were analyzed and compared with respect to vaccination status, risk factors, proneness to acute otitis media etc

CONTACTS AND LOCATIONS:
Overall Officials: Marie Gisselsson Solén, MD, Principal Investigator — ENT Department, Lund University Hospital; Ann Hermansson, MD, PhD, Principal Investigator — ENT Department, Lund University Hospital; Åsa Melhus, MD, PhD, Principal Investigator — Department of Clinical Bacteriology, Uppsala University Hospital
Locations (1):
- ENT Department, Lund University Hospital, Lund, Sweden

REFERENCES:
- [Background] Black S, Shinefield H, Fireman B, Lewis E, Ray P, Hansen JR, Elvin L, Ensor KM, Hackell J, Siber G, Malinoski F, Madore D, Chang I, Kohberger R, Watson W, Austrian R, Edwards K. Efficacy, safety and immunogenicity of heptavalent pneumococcal conjugate vaccine in children. Northern California Kaiser Permanente Vaccine Study Center Group. Pediatr Infect Dis J. 2000 Mar;19(3):187-95. doi: 10.1097/00006454-200003000-00003. PMID 10749457
- [Background] Eskola J, Kilpi T, Palmu A, Jokinen J, Haapakoski J, Herva E, Takala A, Kayhty H, Karma P, Kohberger R, Siber G, Makela PH; Finnish Otitis Media Study Group. Efficacy of a pneumococcal conjugate vaccine against acute otitis media. N Engl J Med. 2001 Feb 8;344(6):403-9. doi: 10.1056/NEJM200102083440602. PMID 11172176
- [Background] Harsten G, Prellner K, Heldrup J, Kalm O, Kornfalt R. Recurrent acute otitis media. A prospective study of children during the first three years of life. Acta Otolaryngol. 1989 Jan-Feb;107(1-2):111-9. doi: 10.3109/00016488909127487. PMID 2929308